CLINICAL TRIAL: NCT03614130
Title: Clinical Performance of a Silicone Hydrogel Following Six Nights of Extended Wear
Brief Title: Clinical Performance of a Silicone Hydrogel Contact Lens Following Six Nights of Extended Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CLL949-C005
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Refractive Errors
Keywords: Contact Lens; Extended Wear; Overnight Wear; Contralateral Wear; Vision Correction
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: In this contralateral study, subjects will be randomized to wear the investigational lens in 1 eye and the control lens in the other eye.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- LID011121 (OD) / Biofinity (OS) (Other): LID011121 contact lens worn in the right eye, with comfilcon A contact lens worn in the left eye, as randomized, for approximately 6 nights of extended (overnight) wear
  Interventions: Device: LID011121 contact lens; Device: Comfilcon A contact lens
- Biofinity (OD) / LID011121 (OS) (Other): Comfilcon A contact lens worn in the right eye, with LID011121 contact lens worn in the left eye, as randomized, for approximately 6 nights of extended (overnight) wear
  Interventions: Device: LID011121 contact lens; Device: Comfilcon A contact lens

INTERVENTIONS:
Device: LID011121 contact lens — Investigational silicone hydrogel contact lens
Device: Comfilcon A contact lens — Commercially available silicone hydrogel contact lens
  Other Names: Biofinity

SUMMARY:
The purpose of this clinical study is to evaluate the on-eye performance of an investigational soft contact lens compared to a commercially available soft contact lens following 1 week of extended wear.

DETAILED DESCRIPTION:
Subjects will be randomized to wear the investigational contact lens in 1 eye and the commercially available contact lens in the other eye. Subjects will be expected to attend 3 scheduled study visits: Day 1 Baseline/Dispense; Day 2 Follow-up; and Week 1 Follow-up/Exit. The expected duration of exposure to each of the study lenses for all randomized, completed subjects was approximately 7 days / 6 nights of wear.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Institutional Review Board/Ethics Committee-approved Informed Consent form.
* Successful wear of spherical soft contact lenses in both eyes during the past 3 months for a minimum of 5 days per week and in an extended wear modality a minimum of 1 night per week.
* Best Corrected Visual Acuity (BCVA) of 20/25 or better in each eye.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any condition, use of medications, or surgery that could contraindicate contact lens wear, as determined by the Investigator.
* Current Biofinity© lens wearer.
* Pregnant or breast-feeding.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (2):
- United States (2):
  - Alcon Investigative Site, Johns Creek, Georgia
  - Alcon Investigative Site, Brentwood, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | LID011121 (OD) / Biofinity (OS) | Biofinity (OD) / LID011121 (OS)
Started | 10; 20 eyes | 12; 24 eyes
Completed | 10; 20 eyes | 12; 24 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All eyes exposed to a study lens evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID011121 (OD) / Biofinity (OS) | Biofinity (OD) / LID011121 (OS) | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (7.7) | 38.3 (10.3) | 40.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA) With Study Lenses, Collected by Eye
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Day 1 Dispense; Day 2 Follow-up (ideally within 4 hours of awakening); Week 1 Follow-up/Exit
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID011121: LID011121 contact lens worn in the right eye or left eye, as randomized, for approximately 6 nights of extended (overnight) wear
- Biofinity: Comfilcon A contact lens worn in the right eye or left eye, as randomized, for approximately 6 nights of extended (overnight) wear
Arm/Group | LID011121 | Biofinity
Number analyzed (Participants) | 22 | 22
Number analyzed (eyes) | 22 | 22
logMAR
  Day 1 Dispense | -0.04 (0.06) | -0.06 (0.06)
  Day 2 Follow-up | -0.06 (0.11) | -0.09 (0.06)
  Week 1 Follow-up/Exit | -0.06 (0.07) | -0.08 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 7 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all eyes exposed to a study lens evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID011121 - Ocular: Events reported in this group occurred while exposed to the LID011121 contact lenses
- Biofinity - Ocular: Events reported in this group occurred while exposed to the comfilcon A contact lenses
- Nonocular/Systemic: Events reported in this group occurred during exposure to the study contact lenses
Arm/Group | Pretreatment | LID011121 - Ocular | Biofinity - Ocular | Nonocular/Systemic
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03614130/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03614130/SAP_001.pdf